CLINICAL TRIAL: NCT07081984
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Immunogenicity of TI-0093 Injection in Patients With Recurrent/Metastatic HPV-16 Positive Solid Tumors
Brief Title: Study of TI-0093 Injection With Recurrent/Metastatic HPV-16 Positive Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Therorna (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0093101
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HPV 16+ Recurrent or Metastatic Cancer; HNSCC; Cervical Cancer
Keywords: Therapeutic tumor vaccine; Circular RNA
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TI-0093 injection (Experimental): Therapeutic tumor vaccine: TI-0093 injection. Different dose levels of TI-0093 injection. Route of administration: Muscle
  Interventions: Biological: therapeutic tumor vaccine

INTERVENTIONS:
Biological: therapeutic tumor vaccine — TI-0093 injection will be administered intramuscularly on Day1, Day8, Day15, Day29 and Day43.

SUMMARY:
This is a phase I, open-label, dose escalation study to assess the safety, tolerability, efficacy and immunogenicity of TI-0093 injection in patients with recurrent or metastatic HPV-16 positive solid tumors.

The primary objectives of the study are to assess safety and tolerability of TI-0093 injection in patients with recurrent or metastatic solid tumors, and to determine the maximum tolerated doses (MTDs) and recommended Phase 2 doses (RP2Ds) of TI-0093 injection.

DETAILED DESCRIPTION:
All potential study candidates will provide informed consent and undergo screening procedures to determine their study eligibility. After a screening period of up to 28 days, qualified patients will be enrolled to receive their assigned dose of TI-0093 injection. Patients will receive a total of five doses of TI-0093 administered muscularly on Day1, Day8, Day15, Day29 and Day43, respectively. Dose-limiting toxicities (DLTs) will be assessed for at least 28 days after the first dose of a given regimen. During the study, patients will be evaluated for safety, toxicity, immunogenicity, ORR, DOR, DCR, and PFS per protocol.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible for participation in this study:

1. The patient provides written informed consent for the study.
2. Willing to comply with the visit plans, treatment plans, and other requirements of the study schedule.
3. Previous HPV16+ solid tumors.
4. 18 to 75 years of age at the time of informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with no deterioration over the previous 2 weeks.
6. Estimated life expectancy of more than 12 weeks.
7. Previous HPV16 positive head and neck, cervical and other carcinoma patients with recurrent or metastatic disease, who have progressed after standard therapies, or for whom no further standard therapies are available.
8. Patients should have at least 1 measurable lesion at baseline according to the definition of RECISTv1.1.
9. Absolute neutrophil count ≥ 1.5 ×10^9/L, without the use of granulocyte colony stimulating factors such as filgrastim within 2 weeks prior to study treatment. Platelet count ≥ 100 × 10^9/L without transfusion within 2 weeks (≤ 14 days) prior to study treatment. Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin within 2 weeks (≤ 14 days) prior to study treatment.
10. Aspartate transaminase and alanine aminotransferase ≤ 3 × upper limit of normal (ULN) (patients with liver metastasis < 5 × ULN), and total bilirubin ≤ 1.5 × ULN (patients with Gilbert's Syndrome ≤ 3 × ULN).
11. Adequate renal function defined by either a creatinine clearance ≥ 45 mL/min (by Cockcroft-Gault formula) or serum creatinine < 1.5 × ULN.
12. Prothrombin time ≤ 1.5 × ULN; activated partial thromboplastin time ≤ 1.5 × ULN; international normalized ratio ≤ 1.5 × ULN.
13. Left ventricular ejection fraction ≥ 50% measured by echocardiogram.
14. Females of childbearing potential and males whose partners are of childbearing potential agree to the use effective contraception from signing informed consent form to 90 days after the last dose of TI-0093 injection. The test results of HCG of females with childbearing potential should be negative within 7 days prior to the first dose of TI-0093 injection.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria cannot be enrolled:

1. History of any therapeutic HPV vaccination. History of any live viral vaccine or attenuated live vaccine therapies within 4 weeks prior to the first dose of TI-0093 injection.
2. History of life-threatening hypersensitivity or known to be allergic to any ingredients contained in the TI-0093 injection.
3. Females who are pregnant or breastfeeding. Patients who plan to donate sperm or eggs from signing informed consent form to 90 days post the last dose of TI-0093 injection.
4. Patients with underlying comorbidity will be excluded:

   A. Active known second malignancy, except for any of the following: basal cell carcinoma, squamous cell skin cancer, in situ cervical cancer and non-muscle invasive bladder cancer, which were recovered from adequate clinical treatment, and other cancers treated by surgery alone whose disease-free survival were 5 years and above.

   B. Meningeal metastases, spinal cord compression or symptomatic brain metastases within 28 days prior to the first dose of TI-0093 injection (except for patients with prior brain metastases who were treated and clinically stable for 4 weeks without corticosteroid or antiepileptic drug treatment).

   C. History of severe pneumonia such as interstitial lung disease within 6 months prior to the first dose of TI-0093 injection.

   D. Major surgery within 4 weeks prior to the first dose of TI-0093 injection. E. Deep vein thrombosis or arterial embolism such as pulmonary embolism within 6 months prior to the first dose of TI-0093 injection.

   F. Active bleeding symptoms or diseases such as active hemoptysis, gastrointestinal bleeding and hemorrhagic gastric ulcer within 28 days prior to the first dose of TI-0093 injection.

   G. Alcohol dependence (averagely more than 2 units of alcohol per day (1 unit = 360 ml of beer, 45 ml of 40% liquor, or 150 ml of wine) which may affect safety assessment judged by the investigator. Drug abuse but unable to quit or mental disorders.

   H. Patients with active autoimmune disease or symptoms that required systemic use of pharmacologic dose of corticosteroid and/or immunosuppressant within 4 weeks prior to the first dose of TI-0093 injection. Exceptions are patients with vitiligo, resolved asthma/atopy, and type 1 diabetes mellitus or hypothyroidism that can be managed by replacement therapy.

   I. Severe or uncontrolled systemic diseases above:
   1. Grade 2 and above myocardial infarction, grade 2 and above myocardial ischemia, or grade 2 and above heart failure based on New York Heart Association (NYHA) classification within 6 months prior to the first dose of TI-0093 injection. Arrhythmia such as QTc ≥ 480ms needs to be treated and uncontrolled hypertension during the screening period.
   2. Any active or uncontrolled infection such as uncontrolled diabetes (defined as HbA1c ≥ 7.5%), asthma, clinically active diverticulitis, abdominal abscess or gastrointestinal obstruction during the screening period.
   3. Active hepatitis B (both hepatitis B virus surface antigen being positive and hepatitis B virus carriers with a viral load > 200 IU/ml), active hepatitis C (both HCV antibody and RNA testing being positive), positive for treponema pallidum in serum or active tuberculosis during the screening period.
   4. Known positive test results for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS). Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.
   5. History of gastrointestinal perforation, gastrointestinal fistula or female reproductive tract fistula within 6 months prior to the first dose of TI-0093 injection. Except for those recovered after treatment judged by the investigator.
   6. Pleural effusion, ascites or pericardial effusion requires puncture aspiration or drainage within 2 weeks prior to the enrollment.
5. Grade 3 and above immune-related AEs or any immune-related AE lead to discontinuation of prior immunotherapy.
6. Any previous AE has not been improved to Grade 1 and below (except for patients with hair loss, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy or other AEs with no safety risk judged by the investigator).
7. Asplenia or insufficiency of spleen function caused by infarct of spleen or thrombosis of splenic vein.
8. Systemic treatment with corticosteroids (≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days prior to the first dose of TI-0093 injection.
9. Washout period for any previous immunomodulatory drugs such as thymosin, interleukin-2, and interferon: last treatment is within 4 weeks prior to prior to the first dose of TI-0093 injection.
10. Washout period for any previous anticancer therapy prior to the first dose of TI-0093 injection:

    1. Last treatment is within 4 weeks for chemotherapy, biologic therapy, target therapy or immunotherapy.
    2. Last treatment is within 2 weeks for radiotherapy, endocrine therapy or oral fluorouracil drugs.
    3. Last treatment is within 7 days for anticancer Chinese medicine.
    4. Last treatment is within 6 weeks for nitrosoureas and mitomycin.
11. Last treatment with investigational product is within 5 half-lives or 4 weeks (which is longer).
12. Any other disease or clinically significant abnormality in laboratory parameters, which in the judgment of the investigator might compromise the safety of the patient or integrity of the study, interfere with the patient participation in the trial or compromise the trial objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment to 28 days post the last dose of TI-0093 injection
  The safety profiles of TI-0093 injection will be assessed in terms of severity, seriousness, frequency of AEs, laboratory results, vital signs, physical examinations, and 12-lead electrocardiogram of the patients enrolled in the study.
DLTs | From enrollment to 3 months.
  DLTs will be assessed for at least 28 days after the first dose TI-0093 injection of a given regimen. Toxicities will be assessed by the National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) v5.0.
RP2D | From enrollment to 3 months.
  The RP2D will be determined based on the observation of MTD.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Confidentiality based on clinical development strategies of TI-0093 injection, IPD sharing will not be planned.